CLINICAL TRIAL: NCT00723749
Title: Post-marketing Surveillance Study (Paper-AWB) for GPs and Clinics: Treatment of Opioid-dependent Patients With SUBOXONE® 2 mg / 8 mg Sublingual Tablets - Acceptability and Safety Data From a Real Life Scenario.
Brief Title: Treatment of Opioid Dependent Patients With Suboxone: Acceptability & Safety Data From Real Life Scenario (Study P05603)
Status: Completed | Type: Observational
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P05603
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2012-04-05 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Opioid-Related Disorders; Opiate Dependence; Drug Abuse
Keywords: Suboxone; Subutex; Buprenorphine; Naloxone
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Suboxone: Patients for whom a drug dependence therapy with SUBOXONE® is planned and indicated, and who have already been pre-treated with SUBUTEX®, or another maintenance drug for at least 6 months.
  Interventions: Drug: Buprenorphine/Naloxone

INTERVENTIONS:
Drug: Buprenorphine/Naloxone — Sublingual combination tablet containing buprenorphine and naloxone at a ration of 4:1, respectively. It is available in two tablet strengths: 2 mg buprenorphine & 0.5 mg naloxone and 8 mg buprenorphine & 2 mg naloxone.
  The only effective and safe use is sublingual administration. SUBOXONE® use will occur on the basis of SPC and is solely aimed at medical-therapeutic necessity.
  Other Names: SCH 000484; SUBOXONE®

SUMMARY:
The aim of this post marketing surveillance study is to investigate the retention rate after 12 months of drug dependence treatment with SUBOXONE® (buprenorphine plus naloxone) of opioid dependent patients under real life conditions.

DETAILED DESCRIPTION:
Nonprobability sampling was done by invitation to volunteer with the intention to document 4 to 5 patients per physician where a substitution therapy with Suboxone is planned and indicated.

ELIGIBILITY:
Inclusion Criteria:

* Both adult and adolescent patients over 15 years of age who have consented to addiction treatment for opioid dependence within the scope of medical, social and psychotherapeutic measures can be included. Therapeutic indications and contraindications for SUBOXONE® must be observed when selecting patients.

Exclusion Criteria:

* In accordance with the product information, it is to be taken into consideration that patients are not suffering simultaneously from acute alcoholism, delirium tremens, or severe respiratory and severe liver insufficiency.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Opioid-dependent patients for whom a drug dependence therapy with SUBOXONE® is planned and indicated, and who have already been pre-treated with SUBUTEX®, or another maintenance drug for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Backmund, PD Dr. med., Principal Investigator — Praxiszentrum im Tal (pit), Munich (Germany)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of sites: Jan - Dec 2008 (General Practitioners, Out-Patient-Clinics, Clinics) Recruitment of patients: Mar 2008 - Dec 2009
Pre-assignment Details: 384 patients were enrolled, 39 datasets were excluded from analysis because 1) physicians withdraw participation agreement, 2) drop-out of patient or final documentation not available
Period: Overall Study
Arm/Group | Suboxone
Started | 345 (384 patients were enrolled, 36 non-eligible datasets were excluded from analysis)
Completed | 182
Not Completed | 163

BASELINE CHARACTERISTICS:
Arm/Group | Suboxone
Number analyzed (Participants) | 345
Age Continuous [Mean (Standard Deviation); unit: years] | 35.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 264
Region of Enrollment [Number; unit: participants]
  Germany | 345

OUTCOME MEASURES:

1. Secondary Outcome: Dosage of SUBOXONE®
Description: Circumstances of switching to SUBOXONE®: Analyse induction and maintenance dose of SUBOXONE®.
Time Frame: Day 1 and Final Assessment (month 12 or time of dropout)
Population: The analysis cohort included all patients prospectively documented, with informed consent, at least 15 years of age at enrollment with written consentment to treatment of drug dependence, for whom SXN-therapy was indicated and planned and with documentation for at least visit 1, visit 2 and visit 12 (end-of-study or discontinuation documentation).
Measure: Mean (Standard Deviation); unit: mg daily dosage of Suboxone
Arm/Group | Suboxone
Number analyzed (Participants) | 345
mg daily dosage of Suboxone
  Dosage: Day 1 | 9.2 (5.1)
  Dosage: Final Assessment | 7.7 (4.4)

2. Primary Outcome: Retention Rate After 12 Months of Treatment With Suboxone
Description: The primary aim of the SUBOXONE® NIS was to document the 12-month retention rate for at least N = 300 subjects with opioid dependence in a real-life scenario in at least N = 70 sites throughout Germany.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Suboxone
Number analyzed (Participants) | 345
% of participants | 59.9 [54.9 to 65.1]

3. Secondary Outcome: Take Home Prescriptions of SUBOXONE®
Description: Circumstances of switching to SUBOXONE®: Analyze if the number of take home prescriptions of SUBOXONE®, reported by the treating physician, increase between day 1 and the final assessment.
  Take Home prescription is defined as a prescription of up to 7 daily dosages SUBOXONE® from the treating physician which allows the patients to receive the prescribed amount of daily dosages SUBOXONE® from a pharmacy to take home and dispense the medication on his own on a daily basis.
  A patient can receive only one take home prescription for up to 7 days at the time.
Time Frame: Day 1 and Final Assessment (month 12 or time of dropout)
Population: as for outcome 1
Measure: Number; unit: participants with take home prescription
Arm/Group | Suboxone
Number analyzed (Participants) | 345
participants with take home prescription
  Frequency: Day 1 | 28
  Frequency: Final Assessment | 82

4. Secondary Outcome: Drug Craving (Subjective Effects of Therapy)
Description: Circumstances of switching to SUBOXONE®: Analyse change of drug craving for opiates by using a 100mm visual analog scale (minimum: 0 = no craving; maximum: 100 = high craving)
Time Frame: Baseline and Final Assessment (month 12 or time of dropout)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Suboxone
Number analyzed (Participants) | 345
Units on a scale
  Craving: Baseline | 32.3 (33.1)
  Craving: Final Assessment | 7.1 (17.2)

ADVERSE EVENTS:
Time Frame: from enrollement (day 0) until 30 days after end of observation = 13 months per patient maximum
Arm/Group | Suboxone
Serious Adverse Events (participants affected / at risk) | 10/384
Other Adverse Events (participants affected / at risk) | 0/384
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Suboxone (N=384)
alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) — C2 withdrawal - termination of treatment
non-compliance (Social circumstances) | 1 (1) — concomitant heroin use
planned abortion (Surgical and medical procedures) | 1/94 (1)
adjustment disorder (Psychiatric disorders) | 1 (1) — hospitilization in psychiatry
alcohol misuse (Psychiatric disorders) | 1 (1)
acute psychosis (Psychiatric disorders) | 1 (1) — acute exacerbation of psychosis
medication addiction (Psychiatric disorders) | 1 (4) — serious withdrawal syndrome, craving, red eyes, no bowel movement, risk of relapse = termination of treatment
hospitalization (Surgical and medical procedures) | 1 (1)
epilepsy (Nervous system disorders) | 1 (1)
accident at home (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial results belong to the Sponsor only, all investigators are not allowed to publish trial results without permission of the Sponsor.